CLINICAL TRIAL: NCT04165954
Title: Treating Phobias Using Emotional Regulation Developed by the Tipi Association
Brief Title: Treating Phobia by a New Emotional Regulation Method (Tipi)
Acronym: RE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Luc Nicon, Education Specialist, Founder of "Tipi", a non-profit French association (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0539
Record Dates: First submitted 2019-11-13; First posted 2019-11-18 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Phobic Fear

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* Background In emotional regulation, the patient remembers an emotional situation, focuses his attention on his physical sensations when he relives a recent emotion, and let evolve his sensations.
* Method Evaluate the relevance of this method by an interventional study, in a pre-post mono group, on patients suffering from phobia.
* Objective The investigators aim to validate the effectiveness of this emotional regulation method and compare its results with that of conventional methods. Sessions are individual and repeated until the disappearance of phobic fear.

The present study may contribute to propose a new possibility to treat phobias in a simple and fast way.

DETAILED DESCRIPTION:
Between 2003 and 2006, the investigators conducted an exploratory, prospective and comparative research study, taking each person as their own control, to evaluate the benefits of the type of emotional regulation developed by the Tipi association on a population suffering from phobias.

- Participants Phobias can be categorized by type, as defined in the DSM IV, the standard reference during the study period (American Psychiatriy Association, 2000) : agoraphobias, social phobias, specific situational phobias (claustrophobia, transport phobia), phobias linked to the natural environment (heights, water, fire), to animals (spiders, snakes, amphibians, tentacled shellfish) and other types of specific phobias (fear of physical contact, being dirtied, contaminated, vomiting), phobia of blood - injections - medical techniques - accidents.

The investigators aim to conduct a prior and systematic verification with each person to confirm that their fears were phobias as defined in the DSM IV (American Psychiatriy Association, 2000). The phobia must be diagnosed by a doctor or psychiatrist. Each people must provide a medical certificate that evidenced the diagnosis in writing.

All people must read an information form on "Understanding your emotions" All participants must have suffered from their phobias for a long time. They have to describe their treatment.

Everybody in the study population have to provide a short-written report on the effects of the session(s) 1 week, 1 month, 3 months and 12 months after the session.

* Intervention (see below)
* Follow-up During the one-year follow-up period, the patient was requested to send a written self-assessment of his situation and the change and/or disappearance of his phobia. If the investigators didn't receive the person's assessment, the investigators followed-up with a mail and a phone call.

ELIGIBILITY:
Inclusion criteria :

* Adult: 18-90 years old
* Adult People with phobic fear in the DSM IV classification
* Phobic people: agoraphobia, with or without panic associated, social phobias and specific phobias. Diagnosis of phobias must be established by the medical world during consultations and explorations. This is systematically checked with the patient to see if the fears come under a phobia as defined in the DSM IV, reference at the time in 2006 (ref DSM IV). The list of phobias classified by type is as follows: animal type or insects; natural environment type (phobias storms, height, water ...); blood type - injection - accident (phobia of seeing blood or an accident or having an injection or any other invasive medical procedure); situational type (fear of specific situations such as public transport, tunnels, bridges, elevators, air travel, driving a car or enclosed areas); another type: afraid to choke, to vomit or contract an illness, fear of falling, and fears about loud noises or disguised characters.
* People accepting regular follow-up until one year after the first session.

Exclusion criteria:

Subject unable to read or/and write

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with a phobic fear listed in the DSM IV classification
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2006-12-01 (Actual); Study Completion 2006-12-30 (Actual)

PRIMARY OUTCOMES:
evolution of phobic fear | Assessment at 3 and 12 month after the first session
  evolution of phobic fear

SECONDARY OUTCOMES:
number of sessions needed for the disappearance of phobic fear | 1 day
  number of sessions needed for the disappearance of phobic fear
adverse reaction rate and description | 1 day
  adverse reaction rate and description
existence of physical and psychological sensations experienced during the sessions and just in the course of | 1 day
  existence of physical and psychological sensations experienced during the sessions and just in the course of
degree of process acceptance for the patient | 1 day
  degree of process acceptance for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Luc Nicon, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC